CLINICAL TRIAL: NCT04527133
Title: An Open Non-comparative Study of the Efficacy and Safety of Aprotinin in Patients Hospitalized With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aviron LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVID-APR-01
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; pneumonia; inpatients
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Aprotinin; gordox

STUDY DESIGN:
Intervention Model Description: A non-comparative study of the efficacy and safety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1/Group 1 (Experimental): Intravenous Aprotinin in addition to standard care: 1 000 000 KIU IV daily during 3 days
  Interventions: Drug: Aprotinin
- Stage 2/Group 2 (Experimental): Inhaled Aprotinin in addition to standard care: 625 KIU 4 times per day during 5 days
  Interventions: Drug: Aprotinin
- Stage 2/Group 3 (Experimental): Intravenous Aprotinin in addition to standard care that includes Favipiravir: 1 000 000 KIU IV daily during 5 days
  Interventions: Drug: Aprotinin

INTERVENTIONS:
Drug: Aprotinin — Intravenous or inhalation
  Other Names: Gordox®

SUMMARY:
The observational study will be carried out in two stages. At the first stage, the efficacy and safety of Aprotinin intravenous infusion as add-on therapy to the standard of care will be studied. At the second stage, two groups will be included: the first group will be the inhaled Aprotinin add-on therapy, the second group will be intravenous Aprotinin in combination with Favipiravir.

DETAILED DESCRIPTION:
Primary objective of the study is to evaluate the efficacy of Aprotinin as add-on therapy in patients hospitalized with COVID-19 using the following parameters:

* The time to elimination of SARS-CoV-2 virus until Day 10;
* The time to C-reactive protein (CRP) normalization until Day 10;
* The time to D-dimer normalization until Day 10.

Secondary objectives are to evaluate the following parameters of efficacy and safety of Aprotinin add-on therapy in patients hospitalized with COVID-19:

* The time to body temperature normalization (<37oC);
* Changes from baseline of the laboratory parameters during 14 days: hematology, CRP, coagulogram;
* Changes of lung injury on CT scan on Day 7 and Day 14 from baseline;
* Frequency of clinical status improvement by 2 scores in accordance with the WHO Ordinal scale of clinical improvement (WHO-OSCI) or discharge from the hospital before Day 14;
* Frequency of transfer to the Intensive Care Unit (ICU), frequency of the non-invasive ventilation, frequency of the invasive ventilation and mortality rate;
* Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) of various severity according to subjective complains, physical examination, vital signs, laboratory tests and ECG.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent Form for participation in the study;
2. Adult male or female ≥18 years of age;
3. Body mass < 90 kg;
4. Positive qualitative RNA SARS-CoV-2 PCR analysis at screening;
5. Score 4 on the WHO-OSCI (added at Stage 2);
6. Subjects with moderate-to-severe disease with the follow conditions and symptoms:

   * Pneumonia;
   * Fever > 38°C;
   * Blood serum CRP > 10 mg/L.
7. Agreement to use medically acceptable forms of birth control during the study (contraceptive with spermicide).

Exclusion Criteria:

1. Severe disease with one of the follow criteria:

   * Respiratory rate > 35 per minute that doesn't decrease after body temperature reducing to normal or subfebrile level;
   * Saturation ≤ 93% at rest;
   * Partial pressure of arterial oxygen (PaO2) < 60 mmHg;
   * Oxygenation index (РаО2/FiO2) ≤ 200 mmHg;
   * Partial pressure of arterial CO2 (PaCO2) > 60 mmHg;
   * Septic shock.
2. Chronic liver and kidney diseases in terminal stage;
3. Other organs failure requiring control and treatment in the ICU;
4. Subjects with HIV;
5. Using of Aprotinin during 6 months prior to screening; hypersensitivity to any of the drug components;
6. Participation in any other clinical trial or using of other study drugs during 28 days prior to screening;
7. Pregnant or lactating women or women planning pregnancy during the clinical study; women with child-bearing potential (including women non-sterilized surgically and in postmenopause for less than 2 years) not using medically acceptable forms of birth control;
8. Inability to read or write; unwillingness to understand and follow the Protocol procedures; non-compliance with the regimen of taking medications or performing procedures that, according to the Investigator, may affect the results of the study or the safety of the patient and prevent the patient from further participation in the study; any other comorbid medical or serious mental conditions that make patient ineligible for participation in the clinical study, limits the ability to obtain informed consent, or may affect patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to elimination of SARS-CoV-2 virus | 10 days
  Time to two negative PCR tests with at least 24 hours interval [days]
Time to CRP normalization | 10 days
  Time to CRP <10 mg/L [days]
Time to D-dimer normalization | 10 days
  Time to D-dimer <243 ng/mL [days]

SECONDARY OUTCOMES:
Time to body temperature normalization | 14 days
  Time to body temperature <37oC [days]
Change in absolute neutrophil count (ANC) | Baseline to Day 14
  Change of ANC [cells/L]
Change in white blood cells (WBC) | Baseline to Day 14
  Change of WBC [cells/L]
Change of CRP | Baseline to Day 14
  Change of CRP [mg/L]
Change of D-dimer | Baseline to Day 14
  Change of D-dimer [ng/mL]
Change in fibrinogen | Baseline to Day 14
  Change of fibrinogen [g/L]
Change of Quick's value | Baseline to Day 14
  Change of Quick's value [%]
Change of international normalized ratio (INR) | Baseline to Day 14
  Change of INR [score]
Changes of lung injury on CT scan | Baseline to Day 14
  Improvement, no change or worsening of the lung injury on CT scan [proportion of patients]
Frequency of clinical status improvement by 2 scores in accordance with the WHO-OSCI or discharge from the hospital | 14 days
  Frequency of clinical status improvement by 2 scores in accordance with the WHO-OSCI or discharge from the hospital [proportion of patients]
Frequency of deterioration of the patients' status | 14 days
  Frequency of transfer to the ICU, non-invasive ventilation, invasive ventilation and mortality rate [proportion of patients]
Frequency of AEs and SAEs | 14 days
  Frequency of AEs and SAEs of various severity according to subjective complains, physical examination, vital signs, laboratory tests and ECG [% of patients]

CONTACTS AND LOCATIONS:
Overall Officials: Elena Simakina, MD, Principal Investigator — Clinical Hospital #1, Smolensk
Locations (1):
- Regional State Budgetary Healthcare Institution "Clinical Hospital №1", Smolensk, Russia

IPD SHARING:
Plan to Share IPD: No
not planned